CLINICAL TRIAL: NCT00968838
Title: Comparative Study of Radiated and Unradiated Leukocyte Transfusions for Patients With Life-threatening Infections: A Collaborative Study by the Leukemia Department and Laboratory Medicine
Brief Title: A Study for Leukemia Patients With Life-Threatening Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-0797
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Leukemia
Keywords: White Blood Cell Transfusion; Radiated Cells; Unradiated Cells; Leukocyte Transfusions; Life-threatening Infections
MeSH Terms: conditions — Leukemia | interventions — Leukocyte Transfusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-radiated White Blood Cell Transfusion (Experimental): Four (4) non-radiated white blood cell transfusions. Each transfusion given daily and taking from 1 hour to several hours depending on toleration of the treatment.
  Interventions: Procedure: White Blood Cell Transfusion
- White Blood Cell Transfusion (Experimental): Four (4) standard white blood cell transfusions (with radiation). Each transfusion given daily and taking from 1 hour to several hours depending on toleration of the treatment.
  Interventions: Procedure: White Blood Cell Transfusion

INTERVENTIONS:
Procedure: White Blood Cell Transfusion — 4 Transfusions, each taking approximately 1 hour:
  Patients <50 years of age receive 4 standard transfusions before they are randomized to receive further radiated or non radiated transfusions.
  Patients >50 years of age are randomized to receive either radiated or non radiated transfusions.

SUMMARY:
The goal of this clinical research study is to compare the effectiveness of a white blood cell transfusion with radiated cells to a white blood cell transfusion with cells that have not been radiated. The safety of this procedure will also be studied.

DETAILED DESCRIPTION:
Radiated White Blood Cell Transfusions:

White blood cell transfusions from a volunteer donor may contain blood cells that your body can react with to produce a disorder called transfusion-associated graft versus host disease. This means that some of the injected white blood cells can reproduce in your body and react with your own tissues and create side effects. To avoid this, the blood is radiated (changed through radiation) to kill all the cells that can divide. But this radiation also may destroy some of the infection-fighting capacity of the white blood cell transfusion, this may decrease the effectiveness of these white blood cell transfusions. Radiating white blood cells is the standard procedure that has been used to treat serious, life-threatening infections.

Non-Radiated White Blood Cell Transfusions:

If the white blood cells are not radiated, it may increase the effectiveness of these white cell transfusions. This may help the white blood cells to make more infection-fighting white blood cells. But, the cells that are also responsible for the transfusion-associated graft versus host disease will not be killed. This increases the risk that you could have this complication.

Study Groups:

If you agree to take part in this study, and if you are one of the first 40 patients, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You or your physician will not know the results of this randomization. If you are in Group 1, you will have a non-radiated white blood cell transfusion. If you are in Group 2, you will have a standard white blood cell transfusion (with radiation). If you are less than 50 years old, you will receive 4 transfusions of radiated white cells. If you continue to show signs and symptoms of infection you will receive additional white cell transfusions based on the group you were randomized to.

If you are after the first 40 patients, you will be placed in a group that the study doctor thinks will most benefit you. It is important to note that this study is designed as a "adaptive randomization" which means that as the outcome for each individual is observed, the next patient receives the product which is most likely to be beneficial and least likely to be harmful.

White Blood Cell Transfusion:

Before the transfusion, a nurse will take your temperature, breathing rate and blood pressure. During the transfusion a nurse will watch you closely. Side effects sometimes occur during and soon after the transfusion. You may be given a drug to help or reduce any side effects.

If you are in Group 2, you will receive 4 standard white blood cell transfusions (with radiation).

If you still have an infection after 4 transfusions and the doctor thinks it is necessary, you will have additional transfusions. You will continue to have transfusions until the doctor feels the infection has been controlled. If you experience graft-versus-host disease (GVHD), this will be up to your doctor's discretion.

If you need a white blood cell transfusion for a new infection or for an infection that comes back, you will receive the same type of transfusion as you received before.

If you were discharged from the hospital and your doctor would like for you to continue receiving white blood cell transfusions, you will be able to receive them as an outpatient.

Each transfusion will take from 1 hour to several hours depending on how you tolerate the treatment. Each transfusion will be given daily or as close to daily as possible.

Before every infusion, blood (about 1 tablespoon) will be drawn to measure the number of white blood cells in your blood.

Length of Study:

You will receive transfusions until your doctor feels the infection has been controlled.

This is an investigational study. White blood cell transfusions are considered standard procedure for the treatment of serious, life threatening infections.

Up to 150 patients will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hematologic malignancy admitted to the Leukemia service.
2. Severe neutropenia defined as Absolute neutrophil count (ANC) less than or equal to 1000.
3. Persistent fever and/or signs of life threatening infection despite 48 hours on antibiotics.
4. Sign a written informed consent form.
5. Greater than 18 years of age.

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emil J Freireich, MD, BS, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 07/16/2008 through 7/14/2011. All participants recruited at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of 178 participants registered, there were 108 participants included in the study and analysis. The 70 participants excluded were ineligible or unable to be matched with a transfusion donor.
Period: Overall Study
Arm/Group | Non-radiated White Blood Cell Transfusion | White Blood Cell Transfusion
Started | 50 | 58
Completed | 50 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-radiated White Blood Cell Transfusion | White Blood Cell Transfusion | Total
Number analyzed (Participants) | 50 | 58 | 108
Age Continuous [Median (Full Range); unit: Years] | 57.5 [20 to 84] | 60 [19 to 79] | 59 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 24 | 33 | 57
Region of Enrollment [Number; unit: participants]
  United States | 50 | 58 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive at Day 30
Description: Participant survival measured over the 30 days subsequent to the first granulocyte transfusion. Collecting complete blood counts (CBCs) pre and post transfusion allows determination of whether the duration of neutrophil replacement differs between the two study groups (comparing unradiated white blood cells to radiated white blood cell infusion).
Time Frame: 30 Days
Measure: Number; unit: Participants
Arm/Group | Non-radiated White Blood Cell Transfusion | White Blood Cell Transfusion
Number analyzed (Participants) | 50 | 58
Participants | 31 | 39

ADVERSE EVENTS:
Time Frame: Participants followed from baseline to minimally 30 days post transfusion(s). Adverse event data collection for all participants was over a study period of 3 years.
Arm/Group | Non-radiated White Blood Cell Transfusion | White Blood Cell Transfusion
Serious Adverse Events (participants affected / at risk) | 5/50 | 3/58
Other Adverse Events (participants affected / at risk) | 3/50 | 2/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-radiated White Blood Cell Transfusion (N=50) | White Blood Cell Transfusion (N=58)
Infection (Infections and infestations) | 4 (4) | 2 (2) — Not treatment related
Disease Progression (General disorders) | 1 (1) | 1 (1) — Disease related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-radiated White Blood Cell Transfusion (N=50) | White Blood Cell Transfusion (N=58)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No